CLINICAL TRIAL: NCT03190837
Title: A Long-term Follow-up Study of Gaucher Disease
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00081246
Record Dates: First submitted 2017-05-26; First posted 2017-06-19 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Gaucher Disease
Keywords: gaucher; gaucher disease
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study aims are to: a) identify the long-term natural history of Gaucher disease, b) evaluate long-term treatment efficacy of enzyme replacement therapy (ERT) and substrate reduction therapy (SRT), and c) identify potential long-term complications of this disorder. These aims will be accomplished through long-term record review of individuals with all three types of Gaucher disease.

DETAILED DESCRIPTION:
The study aims (aims a-c) will be accomplished by the systematic monitoring of health records. Health information will be extracted from medical records for patients followed at Duke. Medical records will be requested from treating physicians outside of Duke. The PI, (Dr. Kishnani) a recognized expert in Gaucher disease, is a consultant to the treating physician of virtually all subjects in this study. Subject health status will be monitored at least on an annual basis and as regularly as the medical information is obtained from the treating physician. Enrollment in this study will not alter the standard of care treatment for patients with Gaucher disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Gaucher Disease

Exclusion Criteria:

* Not meeting Inclusion criteria

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: We will be recruiting patients with Gaucher Disease of all ages, followed at Duke University Medical Center, or non-Duke patients who have contacted Duke and expressed interest in participating.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-06-12 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Document effects of Gaucher disease in different systems of body, including nervous system, liver, and spleen. | 10 years
  Use Gaucher patient's natural histories to understand effects of Gaucher Disease long term.

SECONDARY OUTCOMES:
Document adverse events subjects experience on enzyme replacement therapy | 10 years
  Use Gaucher patient's therapy history to understand effects of enzyme replacement therapy long term.
Document adverse events of subjects on substrate reduction therapy | 10 years
  Use Gaucher patient's therapy history to understand effects of substrate reduction therapy long term.
Document long-term complications in Gaucher Disease. | 10 years
  Use Gaucher patient's natural histories to understand long-term complications of Gaucher Disease.
Change in 36-Item Short Form Survey (SF-36) collected every 6 months/1 year. | 10 years
  We will use the SF-36 that will be collected every 6 months to 1 year to assess quality-of-life in Gaucher patients.
Change in Small Fiber Neuropathy Screening List (SFNSL) collected every 6 months/1 year. | 10 years
  The investigators will use the Small Fiber Neuropathy Screening List every 6 months to 1 year to monitor small fiber neuropathy symptoms in Gaucher patients.
Document number of subjects experiencing neurological symptoms related to Gaucher, by using Neurological Follow-up exam | 10 years
  The investigators will use the Neurological follow-up exam, that will be performed at return visit and every 6 months to 1 year afterward, to screen patients for neurological symptoms related to Gaucher Disease.
Change in Parkinson's checklist collected every 6 months/1 year. | 10 years
  The investigators will use the Parkinson's checklist that will be collected every 6 months to 1 year to screen patients for Parkinson's symptoms potentially related to Gaucher Disease.

CONTACTS AND LOCATIONS:
Overall Officials: Priya Kishnani, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No